CLINICAL TRIAL: NCT02491697
Title: Randomized Controlled Trial Comparing Dendritic Cells Co-cultured With Cytokine-induced Killer Cells Immunotherapy Combined With Capecitabine Versus Capecitabine Monotherapy in Advanced Breast Cancer
Brief Title: Immunotherapy Combined With Capecitabine Versus Capecitabine Monotherapy in Advanced Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First People's Hospital of Changzhou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CZ1H-BC-001
Record Dates: First submitted 2015-07-01; First posted 2015-07-08 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2015-07

CONDITIONS: Breast Cancer
Keywords: DC-CIK; Breast cancer; Capecitabine
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Capecitabine Monotherapy (Active Comparator): Patients with advanced breast cancer accept capecitabine monotherapy.
  Drug: Capecitabine
  Interventions: Drug: Capecitabine Monotherapy
- DC-CIK Immunotherapy+Capecitabine (Experimental): Biological/Vaccine: DC-CIK DC-CIK immunotherapy combined with capecitabine are used to treat advanced breast cancer.
  Drug: Capecitabine
  Interventions: Biological: DC-CIK Immunotherapy; Drug: Capecitabine Monotherapy

INTERVENTIONS:
Biological: DC-CIK Immunotherapy — DC-CIK cells are used to treat advanced breast cancer with capecitabine.
  Other Names: DC-CIK
  Arms: DC-CIK Immunotherapy+Capecitabine
Drug: Capecitabine Monotherapy — All patients receive capecitabine monotherapy (2500 mg/m2 twice daily) for 2 weeks followed by a 1-week rest period.And the treatment is repeated every 3 weeks.
  Other Names: Capecitabine

SUMMARY:
The prognosis of advanced breast cancer does not improve much recently although varies of adjuvant drugs have been tried.Dendritic cells co-cultured with cytokine-induced killer cells(DC-CIK) immunotherapy has been proved to improve survival in several cancers, but its role in advanced breast cancer stains unclear. The purpose of this study is to evaluate the efficacy and safety of DC-CIK immunotherapy combined with capecitabine versus capecitabine monotherapy for the treatment of advanced breast cancer.

DETAILED DESCRIPTION:
1.400 patients with advanced breast cancer should be definitively diagnosis based on histopathology, according to the 7th American Joint Committee on Cancer(AJCC) Cancer Staging Manual.

2.All patients will be randomly divided into group A（DC-CIK immunotherapy combined with capecitabine ) or group B（capecitabine monotherapy).

3.Patients in group A will receive 4 cycles of DC-CIK treatment (every 1 year) and capecitabine(continuous).Patients in group B will receive only capecitabine monotherapy(continuous) .

4.The response is assessed using Response Evaluation Criteria in Solid Tumor Group (RECIST) guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed with advanced breast cancer.
* Eastern Cooperative Oncology Group (ECOG) performance status was 0 - 2.
* Hemoglobin≥10.0g/dL, Neutrophil count≥1.5×10^9/L, Platelet count≥75×10^9/L; total bilirubin(TBIL)≤1.5×ULN; alkaline phosphatase(AKP), aspartate aminotransferase(AST),ALT≤2.5×ULN(without metastasis of the liver), AKP,AST,ALT≤5×ULN(with metastasis of the liver); BUN≤1.5×ULN, Cr≤1.5×ULN.
* Patient received 1-2 kinds of cytotoxic chemotherapy previously.
* Patient never received capecitabine or other oral fluorouracil.

Exclusion Criteria:

* Patients who are suffering from serious organ dysfunction.
* HIV positive or other immunodeficiency disease.
* Patients who had used long time or are using immunosuppressant drugs.
* Patients who had active infection.
* Patients who were allergic to fluorouracil.
* Pregnant or lactating women.
* History of other malignancies.
* Other situations that the researchers considered unsuitable for this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2016-02; Primary Completion 2030-08 (Estimated); Study Completion 2033-08 (Estimated)

PRIMARY OUTCOMES:
Overall Survival(OS) | 1 year

SECONDARY OUTCOMES:
Disease-free survival | 6 months

OTHER OUTCOMES:
Number of participants with side effects | 1 week
  The side effect was evaluated according to WHO standards, including diarrhea, nausea, vomiting, hand-foot syndrome and neutropenia.
Clinical benefit response ( composite) | 2 months
  complete response(CR),partial response(PR),stable disease(SD)and progressive disease(PD).